CLINICAL TRIAL: NCT01080755
Title: Study on the Prescription of the Growth Hormone Saizen® for Adults in France and Follow-up of Treated Patients
Brief Title: Metabolic Endocrinology and Growth Hormone in Adults
Acronym: MEGHA FRANCE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: IMP 24428
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Adult Growth Hormone Deficiency
Keywords: Adult Growth Hormone Deficiency; Pituitary; Saizen; Somatropin; Growth Hormone
MeSH Terms: conditions — Dwarfism, Pituitary; Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicentric, longitudinal, observational study with the prospective follow-up of Adult subjects with Growth Hormone Deficiency (AGHD) being treated with Saizen, every six months in the first year and then annually. At the request of health authorities, the sponsor has arranged for the follow-up of prescriptions and treated subjects within the scope of this indication.

DETAILED DESCRIPTION:
Adult growth hormone deficiency can lead to various effects. In some subjects, an increase is observed in the body fat mass and often, there is an increase in blood lipid levels, which also leads to an increase in risk of death by cardiovascular diseases. Sometimes muscle mass is reduced, thus affecting physical performances, which cannot be rectified by exercise alone. And finally, there is a decline in bone density, which increases the risk of fractures. In general, most of the subjects with inadequate growth hormone secretion also show a deficiency in other hormones secreted by the hypophysis (pituitary gland). In spite of an adequate substitution of the possible related hormonal deficiency, these subjects also present psychomotor retardation, decrease in tonus and vitality, emotional lability, a feeling of social isolation and sexual problems.

In France, marketing approval had been granted to different recombinant growth hormones (GH), including Saizen, for treating AGHD subjects. The indication of Saizen in adults is as follows: marked deficiency in GH documented by a dynamic test indicating somatotroph deficiency. The therapeutic benefits of Saizen as well as its good tolerance has been demonstrated in the marketing approval indications. It has been shown that this treatment results in a significant improvement in the body composition and cardiac function of AGHD subjects.

After receiving the marketing approval for Saizen on the basis of this indication in adults, the sponsor, has set-up a study in France, at the request of health authorities, to ensure a follow-up of the prescriptions and treated subjects in the use of Saizen post marketing approval. This request of the health authorities is also mentioned in the Treatment Information Form.

OBJECTIVES

* To ensure the longitudinal follow-up of GH-deficient adult subjects treated with Saizen in France, with the description:

  1. of the terms and conditions of prescription,
  2. of the demographic and clinical characteristics of subjects,
  3. of subjects' compliance
  4. of product tolerance.

The data collected in this study will concern the demography, medical history, clinical and biological characteristics of the subjects, the terms and conditions of prescription of Saizen, its tolerance and subjects' compliance. The information will be gathered by all hospital endocrinologist (approximately 200 potential prescribing doctors in France). The prescribing doctor shall care for the subjects on account of the treatment and for medical reasons as per his/her regular practice. The period of inclusion of subjects in the cohort is 3 years. The extension of this inclusion period will be discussed with the health authorities during the third year of inclusion. The follow-up period for each subject included will be 5 years. This follow-up will be carried out at regular intervals of 6 months in the first year (2 intermediate visits before 6 months are also available) and then of 12 months in the subsequent years.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects treated with Saizen, irrespective of whether it concerns a first time prescription or a renewal were enrolled in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult subjects treated with Saizen, irrespective of whether it concerns a first time prescription or a renewal were enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2003-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Longitudinal follow up of subjects treated with Saizen | Data to be collected from the start of the follow-up period up to 5 years (every six months in the first year and then annually)
  Demographic data and medical history (date of birth, sex, diagnosis of the hypophyseal pathology and the GH deficit, other hormonal abnormalities, etc.); Clinical and biological data (size, weight, vital signs, body composition, cardiac function, insulin growth factor -1 (IGF1), blood lipids, etc.); Data on the terms and conditions of prescription of the GH (start date, dose, injection cycle, modifications or discontinuation of treatment); Related treatments and Information of the side effects and problems linked to the injection.